CLINICAL TRIAL: NCT06759831
Title: Clinical and Immunological Outcomes of Living and Deceased Donor Transplantation
Acronym: TxBo2022
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TxBo2022
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-10

CONDITIONS: Transplant Recipient (Kidney)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, prospective, single-centre, non-pharmacological observational study.

The primary objective is to investigate the long-term prognosis of the kidney transplant function of different types of donors.

DETAILED DESCRIPTION:
It provides for the systematic collection of clinical information of patients undergoing kidney transplantation from 01/01/2017 until the Ethics Committee approves the study and the Director General of the IRCCS issues the authorisation. Data collection will continue for 9 years after the start of the study.

Patients participating in the prospective part will be treated according to clinical practice, in accordance with the judgement of the physician and the information reported in the Technical Data Sheet of each individual product of any concomitant therapies administered according to clinical practice. There are no additional study-specific visits/examinations for enrolled patients and any data recorded for the purposes of the study is collected for care purposes during the patient's normal course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Kidney transplant recipient from any donor.
* Acquisition of Informed Consent to study participation and data processing.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The medical records of all patients undergoing kidney transplantation performed at the O.U. Nephrology, Dialysis and Transplantation of IRCCS AOUBO from January 2017 until the start of the study will be retrospectively reviewed. After that, all kidney transplant recipients over the next 9 years, performed c/o the U.O. Nephrology, Dialysis and Transplantation of IRCCS AOUBO, will be prospectively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1293 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2033-10-01 (Estimated); Study Completion 2033-10-01 (Estimated)

PRIMARY OUTCOMES:
the functionality of kidney transplantation | 1 month, 6 months, 1 year, 5 years, 10 years
  the functionality of the kidney transplant will be assessed by considering the events of graft failure (return to ESRD, kidney retransplantation), and eGFR change (calculated according to the CKD-EPI formula) at 1 month, 6 months, 1 year, 5 years and 10 years after transplantation. A loss of eGFR of 40% within the first 3 years of follow-up from the baseline visit (at discharge from transplantation) is considered a valid surrogate end-point of ESRD.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgia Comai, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Sant'Orsola University Hospital - Nephrology, Dialysis and Transplant Unit, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No